CLINICAL TRIAL: NCT00112138
Title: Effectiveness and Safety of Gabapentin for the Treatment of Hot Flashes in Menopausal Women: A Randomized Controlled Trial
Brief Title: Gabapentin for the Treatment of Hot Flashes in Menopausal Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: North Toronto Primary Care Research Network (Network)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 03-19; Health Canada: CN 082818
Record Dates: First submitted 2005-05-27; First posted 2005-05-30 (Estimated); Last update posted 2011-05-23 (Estimated); Status verified 2011-05

CONDITIONS: Hot Flashes; Menopause
Keywords: gabapentin; hot flashes or flushes; menopause
MeSH Terms: conditions — Hot Flashes; Blushing | interventions — Gabapentin

INTERVENTIONS:
Drug: gabapentin

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of gabapentin compared to placebo in the treatment of hot flashes in postmenopausal women using a phase III randomized controlled trial.

DETAILED DESCRIPTION:
For women who fear developing breast cancer, those who have contraindications to hormone replacement therapy and those who prefer an alternative treatment, there is presently no standard treatment for hot flashes. Women and health care providers have few options other than hormone replacement therapy as evidenced-based trials of alternatives have not shown many effective options. Many non-hormonal agents have been studied including antidepressants, antihypertensives, vitamin E, soy products, black cohosh, acupuncture, and belladonna and ergotamine combinations. Preliminary studies using the antiseizure medication, gabapentin (Neurontin), has demonstrated a substantial reduction in hot flashes. This agent may provide an effective treatment for hot flashes in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Women with substantial hot flashes defined as reporting at least 14 hot flashes per week.
* Postmenopausal women as defined by the natural cessation of menses for 1 year.
* Aged 45 - 65 years.

Exclusion Criteria:

* Women on hormone replacement therapy.
* Women with a surgically induced menopause (oophorectomy).
* Women on tamoxifen or receiving chemotherapy/radiation therapy or planned antineoplastic chemotherapy/radiation therapy.
* Renal function impairment (serum creatinine greater than the laboratory normal range; or creatinine clearance <30ml/min).
* Use of antidepressants with serotonin reuptake mechanisms and antiseizure medications within the past month.
* Neurologic conditions: seizures, vertigo, and syncope.
* Known hypersensitivity to gabapentin and its components.
* Inability to complete questionnaires for any reason including psychiatric disorders.
* History of a hypothalamic dysfunction.
* Life expectancy less than 6 months.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2004-03; Study Completion 2006-02

PRIMARY OUTCOMES:
Compared to placebo, gabapentin effectiveness in reducing hot flash scores in postmenopausal women

SECONDARY OUTCOMES:
The toxicity profile of gabapentin in this population compared with placebo
The impact of gabapentin on quality of life in this population compared with placebo
Correlation of the Menopause-specific Quality of Life (MENQOL) results with the change in hot flash scores

CONTACTS AND LOCATIONS:
Overall Officials: Debra Butt, MSc MD CCFP, Principal Investigator — North Toronto Primary Care Research Network
Locations (1):
- The Scarborough Hospital, Scarborough Village, Ontario, Canada

REFERENCES:
- [Background] Guttuso T Jr, Kurlan R, McDermott MP, Kieburtz K. Gabapentin's effects on hot flashes in postmenopausal women: a randomized controlled trial. Obstet Gynecol. 2003 Feb;101(2):337-45. doi: 10.1016/s0029-7844(02)02712-6. PMID 12576259